CLINICAL TRIAL: NCT00594880
Title: Antiviral Activity of Peg-IFN-Alpha-2A in Chronic HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Wistar Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Luis Montaner, Protocol Chair / Prinicipal Investigator, The Wistar Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIDS-ES 10401; U01AI065279 (NIH)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: HIV; HIV-1; Pegasys; Peg-IFN-Alpha-2A; Viral Suppression; ART cessation; Immune function; Innate Immunity; Toxicity; Immune-based therapy; Treatment interruption
MeSH Terms: conditions — HIV Infections | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegasys 180 mcg/week (Active Comparator): ART replacement treatment with Pegylated Interferon-alpha 2a, 180 mcg/week sc
  Interventions: Drug: Pegylated Interferon-alpha 2a, 180 mcg/week sc
- Pegasys 90 mcg/week (Active Comparator): ART replacement treatment with Pegylated Interferon-alpha 2a, 90 mcg/week sc
  Interventions: Drug: Pegylated Interferon-alpha 2a, 90 mcg/week sc

INTERVENTIONS:
Drug: Pegylated Interferon-alpha 2a, 180 mcg/week sc — Pegylated Interferon-alpha 2a, 90 mcg/week sc for 24 weeks, 5 weeks in combination with ART, then 7 weeks without ART to primary endpoint (VL < 400 c/ml at 12 weeks) and further 12 weeks without ART (24 weeks) to secondary endpoints
  Other Names: Pegasys
  Arms: Pegasys 180 mcg/week
Drug: Pegylated Interferon-alpha 2a, 90 mcg/week sc — Pegylated Interferon-alpha 2a, 90 mcg/week sc for 24 weeks, 5 weeks in combination with ART, then 7 weeks without ART to primary endpoint (VL < 400 c/ml at 12 weeks) and further 12 weeks without ART (24 weeks) to secondary endpoints
  Other Names: Pegasys
  Arms: Pegasys 90 mcg/week

SUMMARY:
The objective of the study is to compare two different doses of Peg-INF-α-2A (90 or 180 ug/wk) for their ability to maintain viral control when initiated 5 weeks before ART (antiretroviral therapy) interruption in HIV positive, ART-suppressed subjects (viral load <50 copies/ml) as determined by observing the percentages of viral load measurements <400 copies/ml between the two arms over a 24-week period, corresponding to the Pegasys monotherapy period (exclusive of dual ART/Pegasys 5-week period). Primary analysis will be an "intent to treat" analysis and will address the hypothesis that two different doses of Peg-INF-α-2A (90 and 180 ug/week) will be similarly effective at inhibiting viral replication.

DETAILED DESCRIPTION:
The high toxicity of current Anti-Retroviral Therapy (ART) regimens has driven a number of studies investigating therapeutic approaches aimed at reducing drug exposure while maintaining the beneficial effects of immune reconstitution. Preliminary observations in HCV/HIV co-infected individuals already support an antiviral effect by Pegylated Interferon-Alpha-2A (Peg-IFN-Alpha-2A:Pegasys®) on HIV-1 replication; however, the ability of Peg-IFN-Alpha-2A (as a single agent) to maintain long-term suppression of HIV-1 replication in patients who interrupt ART after having achieved immune reconstitution remains undetermined. The rationale for addressing two doses of Peg-IFN-Alpha-2A (180 and 90 ug/week) is based on the antiviral activity reported with both doses and the lower incidence of adverse events associated with doses lower than that approved for HCV therapy (90 versus 180ug/week).

The long-range goal of this proposal is to determine if Peg-IFN-Alpha-2A monotherapy can sustain HIV-1 suppression in the absence of ART in infected individuals. Our short-range goal is to determine the safety, viral suppressive potential and immune correlates of Peg-IFN-Alpha-2A administered upon the cessation of suppressive ART.

Based on the current literature and our preliminary studies, we hypothesize that weekly doses of 90 or 180 ug/wk of Peg-IFN-Alpha-2A administered to pharmacologically-suppressed HIV-infected individuals in the course of antiretroviral therapy (ART) discontinuation will result in equivalent frequency of viral control, with the lower dose resulting in measurably lower rate and intensity of therapy-related adverse events (AE).

We propose to compare two different doses of Peg-IFN-Alpha-2A (90 or 180 ug/wk) as a simplification step to ART, for their ability to maintain viral load suppression when initiated 5 weeks before ART interruption in HIV-infected, ART-suppressed patients (VL<50 copies/ml). Briefly, control will be determined by the the percentages of viral load measurements <400 copies/ml between the two arms over a period of 24 weeks, corresponding to the Pegasys monotherapy period (exclusive of dual ART/Pegasys 5-week period). A threshold of 400 is used based on the known potential for blipping on ART between 50 and 400 copies/ml with no clinical consequence to sustained suppression thereafter (JAMA 2005, 293:817-829). Primary analysis will be an "intent to treat" analysis and will address the hypothesis that two different doses of Peg-IFN-Alpha-2A (90 and 180 ug/week) will be similarly effective at inhibiting viral replication.

The secondary objectives of the research are:

1. To prospectively evaluate dose-dependent, treatment-associated toxicity, safety and tolerability of 29 weekly doses of Peg-IFN-Alpha-2A at 180 ug or 90 ug/week (in association with ART for the initial 5 weeks, followed by 24 weeks of Peg-IFN-Alpha-2A in the absence of ART).
2. To determine innate immunity outcomes correlated to Peg-IFN-Alpha-2A dose and antiviral activity by monitoring Natural Killer (NK) and Dendritic cell (DC) subsets changes and the ability to maintain innate immune function (DC secretory responses, NK antiviral cytotoxic responses)
3. To determine adaptive immunity outcomes correlated to Peg-IFN-Alpha-2A dose and antiviral activity by monitoring T-cell subsets changes and the ability to maintain cell-mediated proliferative and cytokine responses against recall antigens (anti-HIV-1 gag p55).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 but <65 years
* Able and willing to provide informed consent.
* HIV-1 infection documented by any licensed enzyme-linked immunosorbent assay (ELISA) test kit and confirmed by Western Blot at any time prior to or at study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test
* HIV RNA < 75 copies/ml on a regimen of a) 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs) and 1 non-nucleoside RTI (NNRTI) OR b) 2 NRTIs and Protease Inhibitor (PI) for at least 24 weeks OR c) 3 NRTIs
* HIV RNA < 75 copies/ml at screening
* > 6 months ≥ 400 CD4+ T cells/mm3 (CD4 nadir ≥ 200 cells)
* Female subjects with childbearing potential: negative pregnancy test (Beta human horionic gonadotropin (HCG)). Must agree to use appropriate contraceptive methods (barrier devices such as diaphragms or condoms + spermicidal or intrauterine device (IUD) or oral contraceptives) while on study.
* Karnofsky performance scale score of 80% or better
* Willing to adhere to the treatment and schedule approved by the study investigators in conjunction with the patient's primary provider.
* Willing to abstain from immunomodulatory drugs during the study period, with the exception of the study drug (Pegasys®).
* Patient Health Questionnaire (PHQ)-2 score < 2, OR PHQ-9 score< 10, OR PHQ-9 score 10-14 AND medical provider's favorable opinion. In either case, score for PHQ-9 question # 9 (suicidal ideation) must be 0.
* Thyroid stimulating hormone (TSH) within normal range, unless accompanied by thyroid profile consistent with normal thyroid function
* A negative cardiac stress test if >45yrs men/>55yrs women years of age or if below these years of age but with two added risk factors for coronary artery disease [smoking, hypertension (BP >140/90 or on antihypertensive medications), low Hight density lipoprotein (HDL)-associated cholesterol (<40 mg/dL), family history of premature Coronary heart disease (CHD) (<55 yrs males/<65 females)] or a Framingham score > 15% (men) or 10% (women))

Exclusion Criteria:

* Currently pregnant or breast feeding.
* CD4 cell count < 400 or recorded CD4 nadir < 200 cells/mm3
* History of immunomodulatory therapy for over 2 weeks during the 6 months prior to enrollment, including, but not limited to: IFN-Alpha or Beta (recombinant or pegylated), systemic corticosteroids; systemic cancer chemotherapy/irradiation; cyclosporin; tacrolimus (FK-506); OKT-3; any Interleukin, including IL-2; cyclophosphamide; methotrexate; IVIG (gamma globulin); G/M-CSF; hydroxyurea; thalidomide; pentoxifylline; thymopentin; thymosin; dithiocarbonate; polyribonucleoside.
* Significant co-existing medical conditions including: Anemia (Hgb <9.1 men, <8.9 women), Neutropenia (ANC < 1000), Thrombocytopenia (platelet count <50K), Liver disease (AST/ALT > 5x, Total Bilirubin > 1.5x upper limits of normal, or Total Bilirubin >3x upper limit of the norm (ULN) if receiving indinavir), Renal disease (creatinine > 2x upper normal limits), or other conditions, such as active drug/alcohol abuse or dependence which would interfere with study compliance.
* Any history of heart attacks, myocardial infarction or coronary arterial disease (MI/CAD). .
* Prior history of major depression or other severe psychiatric disorder/condition requiring treatment and/or hospitalization
* PHQ-9 score >14, OR PHQ-9 score > 10 - 14 and lack of medical provider's favorable opinion, or score for PHQ-9 answer # 9 (suicidal ideation) > 0.
* Evidence of chronic active Hepatitis B infection (Surface Antigen HBsAg) or Hepatitis C plymerase chain reaction (PCR) positivity at screening (cleared of HCV at entry >6 months).
* Past evidence of medical conditions associated with chronic liver disease including genetic hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures etc.
* History of neutropenia or other hematological abnormalities
* Type I diabetes mellitus, or type II diabetes mellitus that is not controlled with oral agents and/or insulin.
* Ongoing treatment with Isoniazide, Pyrazinamide, Rifabutin, Rifampicin, Diadenosine Ganciclovir, Valganciclovir, Oxymetholone, Thalidomide or Theophylline.
* History of autoimmune processes including Crohn's disease, ulcerative colitis, severe psoriasis, rheumatoid arthritis, myositis, hepatitis etc.
* History of major organ transplantation with an existing functional graft.
* Active coronary artery disease within 24 weeks prior to study
* Hemoglobinopathies such as sickle cell anemia or Thalassemia major.
* Hypersensitivity to Pegasys®or any of its components.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Montaner, DVM, PhD, Study Chair — The Wistar Institute; Jay Kostman, MD, Principal Investigator — Penn-Presbyterian Medical Center; Pablo Tebas, MD, Principal Investigator — University of Pennsylvania; Jeffrey Jacobson, MD, Principal Investigator — Drexel University College of Medicine; Karam Mounzer, MD, Principal Investigator — Jonathan Lax Immune Disorders Clinic- Philadelphia FIGHT
Locations (5):
- United States (5):
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn-Presbyterian Medical Center, Philadelphia, Pennsylvania
  - The Wistar Institute, Philadelphia, Pennsylvania
  - Jonathan Lax Immune Disorders Clinic, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Azzoni L, Foulkes AS, Papasavvas E, Mexas AM, Lynn KM, Mounzer K, Tebas P, Jacobson JM, Frank I, Busch MP, Deeks SG, Carrington M, O'Doherty U, Kostman J, Montaner LJ. Pegylated Interferon alfa-2a monotherapy results in suppression of HIV type 1 replication and decreased cell-associated HIV DNA integration. J Infect Dis. 2013 Jan 15;207(2):213-22. doi: 10.1093/infdis/jis663. Epub 2012 Oct 26. PMID 23105144
- [Derived] Papasavvas E, Azzoni L, Ross BN, Fair M, Howell BJ, Hazuda DJ, Mounzer K, Kostman JR, Tebas P, Montaner LJ. Comparable HIV suppression by pegylated-IFN-alpha2a or pegylated-IFN-alpha2b during a 4-week analytical treatment interruption. AIDS. 2021 Oct 1;35(12):2051-2054. doi: 10.1097/QAD.0000000000002961. PMID 34049356
- [Derived] Chitre AS, Kattah MG, Rosli YY, Pao M, Deswal M, Deeks SG, Hunt PW, Abdel-Mohsen M, Montaner LJ, Kim CC, Ma A, Somsouk M, McCune JM. A20 upregulation during treated HIV disease is associated with intestinal epithelial cell recovery and function. PLoS Pathog. 2018 Mar 5;14(3):e1006806. doi: 10.1371/journal.ppat.1006806. eCollection 2018 Mar. PMID 29505600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: locations: medical clinics (Hospital of the University of Pennsylvania, Jonathan Lax clinic, Drexel University Hospital) Recruitment period: may 8, 2008 to May 27, 2010
Pre-assignment Details: subjects were randomized to the pegasys dose of 180 or 90 mcg/week four weeks after enrollment (week 0: eligibility determination; week 4: enrollment; week 8: randomization and treatment initiation; week 13: ART interruption; week 25: primary endpoint; week 37: secondary endpoints)
Groups:
- Pegasys 180 mcg/Week: ART replacement treatment with Pegylated Interferon-alpha 2a, 180 mcg/week sc
  Pegylated Interferon-alpha 2a, 180 mcg/week sc : Pegylated Interferon-alpha 2a, 90 mcg/week sc for 24 weeks, 5 weeks in combination with ART, then 7 weeks without ART to primary endpoint (VL < 400 c/ml at 12 weeks) and further 12 weeks without ART (24 weeks) to secondary endpoints
- Pegasys 90 mcg/Week: ART replacement treatment with Pegylated Interferon-alpha 2a, 90 mcg/week sc
  Pegylated Interferon-alpha 2a, 90 mcg/week sc : Pegylated Interferon-alpha 2a, 90 mcg/week sc for 24 weeks, 5 weeks in combination with ART, then 7 weeks without ART to primary endpoint (VL < 400 c/ml at 12 weeks) and further 12 weeks without ART (24 weeks) to secondary endpoints
Period: Overall Study
Arm/Group | Pegasys 180 mcg/Week | Pegasys 90 mcg/Week
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegasys 180 mcg/Week | Pegasys 90 mcg/Week | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 45.5 [42.8 to 48.5] | 44 [32 to 49.5] | 45 [40.5 to 49.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: HIV Viral Load < 400 Copies/ml
Description: % of individuals maintaining viral suppression (VL < 400 copies/ml) as compared to the anticipated rate of viral suppression in individuals interrupting ART without interferon (9%)
Time Frame: 12 weeks
Population: excluded 2 withdrawal of consent and 1 lost to follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Pegasys 180 mcg/Week | Pegasys 90 mcg/Week
Number analyzed (Participants) | 10 | 10
percentage of participants | 40 | 50

2. Secondary Outcome: HIV Viral Load < 48 Copies/ml
Description: % of individuals maintaining VL < 48 copies/ml while on pegylated interferon alpha-2a treatment without ART
Time Frame: 12 weeks
Population: % of subjects maintaining VL < 48 copies/ml after 12 weeks of treatment
Measure: Number; unit: percentage of participants
Groups:
- 180 mcg/Week: Patients receiving 180 micrograms/week of pegylated interferon alpha-2a
- 90 mcg/Week: Patients receiving 90 micrograms/week of pegylated interferon alpha-2a
Arm/Group | 180 mcg/Week | 90 mcg/Week
Number analyzed (Participants) | 10 | 10
percentage of participants | 10 | 30

3. Secondary Outcome: HIV Viral Load < 400 Copies/ml
Description: as for outcome 1
Time Frame: 24 weeks
Population: percent of consenting eligible participants (n=8) with VL < 400 at week 24 of treatment
Measure: Number; unit: percentage of eligible participants
Groups:
- 180 mcg/Week: Arm 1 subjects with VL < 400 at week 12 of treatment who elected to continue study treatment for an additional 12 weeks
- 90 mcg/Week: Arm 2 subjects with VL < 400 at week 12 of treatment who elected to continue study treatment for an additional 12 weeks
Arm/Group | 180 mcg/Week | 90 mcg/Week
Number analyzed (Participants) | 3 | 5
percentage of eligible participants | 67 | 80

ADVERSE EVENTS:
Arm/Group | Pegasys 180 mcg/Week | Pegasys 90 mcg/Week
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegasys 180 mcg/Week (N=12) | Pegasys 90 mcg/Week (N=11)
depression (Psychiatric disorders) | 1 (1) | 2 (2) — based on PHQ2/9 questionnaire self evaluatiuon
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Liver toxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) — elevated ALT (grade 3 ACTG)

LIMITATIONS AND CAVEATS:
The follwing limitations of this study should be noted:

* Small number of participants enrolled
* Lack of a control arm interrupting ART without immunotherapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No